CLINICAL TRIAL: NCT02329470
Title: Arterial Stiffness and Blood Pressure Changes After Continuous Positive Airway Pressure (CPAP) Withdrawal for Obstructive Sleep Apnea
Brief Title: Cardiovascular Effects After CPAP Withdrawal for Obstructive Sleep Apnea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Umeå University (Other)
Responsible Party: Principal Investigator, Karl A Franklin, Ass Prof, Umeå University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Dnr: 2010-329-31M
Record Dates: First submitted 2014-12-12; First posted 2014-12-31 (Estimated); Last update posted 2023-03-03 (Actual); Status verified 2023-02

CONDITIONS: Obstructive Sleep Apnea; Cardiovascular Disease
MeSH Terms: conditions — Sleep Apnea, Obstructive; Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- No device, n=50 (Experimental): Withdrawal of device, continuous positive airway pressure treatment during 5 nights
  Interventions: Procedure: Withdrawal of continuous positive airway pressure treatment
- Continue using device, continuous positive airway pressure treatment n=50 (No Intervention): Control group, Continue with device, continuous positive airway pressure treatment

INTERVENTIONS:
Procedure: Withdrawal of continuous positive airway pressure treatment — Withdrawal of continuous positive airway pressure treatment
  Arms: No device, n=50

SUMMARY:
Background: Patients with obstructive sleep apnea run an increased risk of cardiovascular disease including hypertension. Continuous positive airway pressure (CPAP) is the first line of treatment. However, many patients skip CPAP for some nights.

Aims: The primary aim was to investigate the cardiovascular effects of short-term CPAP withdrawal for five nights because of obstructive sleep apnea.

Design: Randomized, parallel controlled trial Inclusion criteria: 100 patients with successful CPAP treatment for moderate to severe obstructive sleep apnea.

Exclusion criteria: Dementia, heart infarction within 3 months, apnea hypopnea index > 10 with CPAP treatment.

Randomization: 50 patients are randomized to sleep 5 days without CPAP and 50 patients to continue with CPAP treatment during the trial.

Primary outcomes: Arterial stiffness, 24-hour blood pressure. Secondary outcomes: Effects of gender on outcome. Effects on brain natriuretic peptide, apnea-hypopnea index, oxygen desaturation-index, urine-catecholamines, blood lipids, C-reactive protein, glucose metabolism (S-glc, HBA1c), insulin resistance, serum creatinine, hemoglobin, daytime sleepiness (ESS, KSS), lung function (FVC, FEV1), airway inflammation (exhaled NO) Procedures: Sleep apnea investigation while patients are treated with CPAP for one night. Urinary samplings during the same night. They are also investigated with 24 h blood pressure measurements. Blood samples are taking fasting in the morning followed by measuring the arterial stiffness (Vicorder, Skidmore Medical UK) including pulse wave analysis using sphygmomanometer (Omron Japan). The same investigations are done at follow-up 5 days later where half of the patients have continued using CPAP treatment and half of them has slept without CPAP.

DETAILED DESCRIPTION:
Patients fulfilling inclusion criteria are invited to the trial after informed consent for baseline and follow-up investigations.

Baseline investigations Day 1 Patients are given a questionnaire. They are given blood pressure monitoring, (ABPM Medical 90217 ambulatory blood pressure monitor, Spacelab) for 24 hours a starting at 8-9 AM. They are also given sleep apnea recorder (Embletta, X 10 system, Embla systems, ResMed) for ambulatory use during the following night, and a container for urinary sampling during the night (urine norepinephrine).

Day 2 Fasting on arrival. Return of the 24-h blood pressure recorder, the sleep apnea recorder and the urine sampling container.

Blood samples at 08.15 am after resting for 15 minutes. Arterial stiffness is measured using arterial pulse wave velocity, radial artery applanation tonometry and office blood pressure. After resting, the measurements starts at 8.30 AM in a room with a temperature of 24°C. Pulse wave velocity (Vicorder, Skidmore Medical, Bristol, UK) is measured in the supine position. The augmentation index is derived from pulse wave analysis obtained from radial artery applanation tonometry on the right arm (SphygmoCor, AtCor Medical, Sydney, Australia).

Lung function and exhaled NO measurements, ECG. Breakfast at around 10.00 am. CPAP time counter check Patients are then randomized with a ration of 1:1 to continue with CPAP or not for the following 5 nights.

Follow-up measurements Day 6 They are given blood pressure monitoring, (ABPM Medical 90217 ambulatory blood pressure monitor, Spacelab) for 24 hours a starting at 8-9 AM. They are also given sleep apnea recorder (Embletta, X 10 system, Embla systems, ResMed) for ambulatory use during the following night, and a container for urinary sampling during the night (urine norepinephrine).

Day 7 Fasting on arrival. CPAP time counter check Return of the 24-h blood pressure recorder, the sleep apnea recorder and the urine sampling container.

Blood samples at 08.15 am after resting for 15 minutes. Arterial stiffness is measured using arterial pulse wave velocity, radial artery applanation tonometry and office blood pressure. After resting, the measurements starts at 8.30 AM in a room with a temperature of 24°C. Pulse wave velocity (Vicorder, Skidmore Medical, Bristol, UK) is measured in the supine position. The augmentation index is derived from pulse wave analysis obtained from radial artery applanation tonometry on the right arm (SphygmoCor, AtCor Medical, Sydney, Australia).

Lung function and exhaled NO measurements, ECG. Breakfast at around 10.00 am. Trials ends and patients are told to continue with CPAP as usual.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older,
* given the written consent to participate in the study,
* 2 months to 2 years of continuous positive airway pressure (CPAP) treatments with good compliance (mean CPAP use of >4 hours/night) during the last month before inclusion
* moderate sleep apnea with Apnea Hypopnea Index >15 before treatment

Exclusion Criteria:

* Apnea hypopnea index > 10 with CPAP treatment,
* heart infarction within 3 months prior to study participation,
* severe dementia,
* determined by study personal having psychological or physical hinder to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2014-12-18 (Actual); Primary Completion 2016-08-31 (Actual); Study Completion 2016-08-31 (Actual)

PRIMARY OUTCOMES:
Arterial stiffness. | 5 days
  Arterial stiffness measured with Vicorder and pulse wave analysis
Systolic and diastolic blood pressure | 5 days
  24 hour blood pressure measurements

SECONDARY OUTCOMES:
Gender differences | 5 days
  Effect of gender on outcomes
Effect on myocardial function | 5 days
  Brain natriuretic peptide
Impact on apnea hypopnea index | 5 days
  apnea-hypopnea index
Effect on oxygen saturation | 5 days
  Oxygen desaturation index
Effect on catecholamines | 5 days
  measurements of urinary catecholamines during one day
Effect on blood lipids in the form triglycerides | 5 days
  serum triglycerides
Effect on blood lipids in the form of cholesterol | 5 days
  serum cholesterol
Effect on systemic inflammation. | 5 days
  C reactive protein (CRP)
Effect on glucose metabolism in the form of fasting glucose | 5 days
  Serum glucose obtained fasting in the morning
Long-term effect on glucose metabolism | 5 days
  serum HbA1c
Glucose metabolism in the form om Insulin levels | 5 days
  fasting serum insulin obtained in the morning.
Effect on renal function | 5 days
  serum creatinine
Effect on hemoglobin | 5 days
  serum hemoglobin
Assessment of daytime sleepiness for a past period of time | 5 days
  Epworth sleepiness scale
Daytime sleepiness assessed at a certain time point | 5 days
  Karolinska sleepiness scale
Effect on lung volumes | 5 days
  Vital capacity
Effect on airway obstructions | 5 days
  Forced vital capacity in one second
Effect on airway inflammation | 5 days
  Exhaled nitric oxide test

CONTACTS AND LOCATIONS:
Overall Officials: Karl A Franklin, Prof, MD, Principal Investigator — umea University; Carin Sahlin, PhD, Study Director — Umea University
Locations (1):
- Dept of Respiratory Medicine, Umeå, Sweden

DOCUMENTS (1):
  • Study Protocol (2013-10-01): https://cdn.clinicaltrials.gov/large-docs/70/NCT02329470/Prot_000.pdf